CLINICAL TRIAL: NCT06143098
Title: Some Hematological Profile in Children With Chronic Kidney Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zeinab Othman AbdelGaleel, principal investigator, Assiut University
Other Study IDs: hematological profile in CKD
Record Dates: First submitted 2023-11-14; First posted 2023-11-22 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: CKD; Hematological Disease
Keywords: CBC in CKD; Iron profile in CKD; Coagulation profile in CKD
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is asses the hematological changes in children with chronic kidney disease stage 3 to 5 including

* Complete blood picture
* Coagulation profile (PT, PC, PTT)
* Iron study

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a major public health issue with an increasing incidence and prevalence worldwide. In CKD, hematological parameters are influenced, it is associated with high morbidity and mortality rates, but there have been very few studies on the hematological profile of children with chronic kidney disease, on follow-up in general, and particularly among chronic kidney disease patients(Melaku.,et al 2022).

CKD is defined by the presence of kidney damage or an estimated glomerular filtration rate (eGFR) less than 60 ml/min/1.73 m2, it can last for 3 months or longer, regardless of the cause. Chronic kidney disease (CKD) is recognized as a major non-communicable disease in children. (Inker.,et al2014).

CKD is classifies it into 6 categories based on glomerular filtration rate (G1 to G5 with G3 split into 3a and 3b). It also includes the staging based on three levels of albuminuria (A1, A2, and A3), with each stage of CKD being sub-categorized according to the urinary albumin-creatinine ratio in (mg/gm) or (mg/mmol) in an early morning "spot" urine sample.( Inker,.et al 2012)

The 6 categories include:

* G1: GFR 90 ml/min per 1.73 m2 and above
* G2: GFR 60 to 89 ml/min per 1.73 m2
* G3a: GFR 45 to 59 ml/min per 1.73 m2
* G3b: GFR 30 to 44 ml/min per 1.73 m2
* G4: GFR 15 to 29 ml/min per 1.73 m2
* G5: GFR less than 15 ml/min per 1.73 m2 or treatment by dialysis The three levels of albuminuria include an albumin-creatinine ratio (ACR)
* A1: ACR less than 30 mg/gm (less than 3.4 mg/mmol)
* A2: ACR 30 to 299 mg/gm (3.4 to 34 mg/mmol)
* A3: ACR greater than 300 mg/gm (greater than 34 mg/mmol). (Inker.,et al2014). hematological parameters such as white blood cell (WBC) include total leukocyte and differential counts, platelet (PLT), and red blood cell (RBC). Parameters, Kidney function ,electrolytes such as Na,k,ca and liver function bleeding time, and pro-thrombin time, are usually affected in CKD . These are common in CKD due to erythropoietin deciency and other factors such as increased hemolysis, suppression of bone marrow erythropoiesis, hematuria, and gastro intestinal blood loss. (George.,et al2015).

All CKD patients, particularly those with an estimated GFR (eGFR) < 60 mL/min/1.73 m2, should be screened for anemia on initial evaluation for CKD. Anemia is defined as Hb < 13 g/dL in men and Hb < 12 g/dL in women, according to WHO criteria. (Hira Shaikh.,et al 2023).

the primary cause of anemia in patients with CKD is insufficient production of erythropoietin by the diseased kidneys. Other factors include iron, folate & B12 deficiency due to nutritional insufficiency or increased blood loss (Hira Shaikh.,et al 2023). acute and chronic inflammation with impaired iron utilization, sever hyperparathyroidism with consequent bone marrow fibrosis and shortened red cell survival in the uremic environment, bleeding due to dysfunctional platelets, and rarely blood loss from hemodialysis(Hira Shaikh.,et al 2023).

Criteria used to define iron deficiency are different among CKD compared to normal renal function. Among CKD patients, absolut iron deficiency is defined when the transferrin saturation (TSAT) is ≤20% and the serum ferritin concentration is ≤100 ng/mL among predialysis and peritoneal dialysis patients or ≤200 ng/mL among hemodialysis patients. Functional iron deficiency, also known as iron-restricted erythropoiesis, is characterized by TSAT ≤20% and elevated ferritin levels. (TSAT = plasma iron divided by the total iron-binding capacity × 100)( Cappellini .,et al 2017) .

untreated prolonged anemia leads to a number of physiologic disorders, including: cardiovascular complications like decreased tissue oxygenation, increased cardiac output, ventricular dilatation and ventricular hypertrophy and increased mortality and morbidity.( Dwijen Das ., et al 2015).

Iron supplementation is recommended for all CKD patients with anemia. There is general agreement according to guidelines that intravenous (i.v.) iron supplementation is the preferred method for CKD patients on dialysis (CKD stage 5D) and either i.v. or oral iron is recommended for patients with CKD(Tolkien.,et al 2015)

ELIGIBILITY:
Inclusion Criteria:

* Childen aged 1:18 years with chronic kidney disease stage 3 to 5 (estimated glomerular filteration rate >60 ml/min per 1.73 m2).

Exclusion Criteria:

* Children >1year.
* Children with chronic kidney disease in stage 1 and 2.
* Children with liver disease.
* Children known blood disorder rather than anemia.
* Children with malignancy.
* Children with recent bleeding tendancy.

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Childen aged 1:18 years with chronic kidney disease stage 3 to 5 (estimated glomerular filteration rate >60 ml/min per 1.73 m2).
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
descreption and observation in Complete blood count parameters in children with CKD | baseline
  asses changes in Complete blood count parameter in children with chronic kidney disease stage 3 to 5
descreption and observation in iron profile in children with CKD | baseline
  asses changes in serum ferritin ,serum iron, Trans ferritin saturation and Total iron binding capacity in children with chronic kidney disease stage 3 to 5
descreption and observation in coagulation profile in children with CKD | baseline
  asses changes in prothrombin time, prothrombin concentration, partial thromboplastin time,and international normalized ratio in children with chronic kidney disease stage 3 to 5

CONTACTS AND LOCATIONS:
Overall Officials: Kotb Abbass, professor, Study Director — Assiut University; Asmaa Ahmed, lecture, Study Director — Assiut University

REFERENCES:
- [Background] Hashmi MF, Shaikh H, Rout P. Anemia of Chronic Kidney Disease. 2024 Jul 23. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK539871/ PMID 30969693